CLINICAL TRIAL: NCT06956547
Title: ResQ117EX-ALC: Expanded Access Use of Nogapendekin-alfa Inbakicept in the Reversal and Maintenance of Absolute Lymphocyte Count (ALC) for the Treatment of Lymphopenia Induced by Chemotherapy, Immunotherapy, and/or Radiation Therapy
Brief Title: Expanded Access Use of Nogapendekin-alfa Inbakicept in the Reversal and Maintenance of Absolute Lymphocyte Count (ALC) for the Treatment of Lymphopenia Induced by Chemotherapy, Immunotherapy, and/or Radiation Therapy
Status: Available | Type: Expanded Access
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ResQ117EX-ALC
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Lymphopenia
Keywords: lymphopenia; lymphopenia induced by chemotherapy; lymphopenia induced by radiation therapy; lymphopenia induced by immunotherapy; absolute lymphocyte count
MeSH Terms: conditions — Lymphopenia | interventions — ALT-803

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: nogapendekin-alfa inbakicept — 1.0mg nogapendekin-alfa inbakicept (NAI) administered by subcutaneous injection no less than every 3 weeks and no more frequently than every 2 weeks between doses in combination with the standard of care schedule of chemotherapy, immunotherapy, and/or radiation therapy. Patients who are known HIV+ will be dosed with NAI at 0.5 mg
  Other Names: NAI; N-803

SUMMARY:
This is a protocol for expanded access use of nogapendekin-alfa inbakicept (NAI) in participants with lymphopenia induced by chemotherapy, immunotherapy, and/or radiation therapy who may benefit from its use, and who are ineligible to participate in a clinical trial using NAI. The primary objective of this protocol is to evaluate the reversal and maintenance of absolute lymphocyte count (ALC) with NAI.

DETAILED DESCRIPTION:
It is now well established that patients undergoing standard of care chemotherapy, immunotherapy, and/or radiation therapy sustain the adverse effects of these agents with a reduction in lymphocyte count (lymphopenia), and a significant clinical effect of reduced overall survival across all tumor types. Severe lymphopenia is defined as absolute lymphocyte count (ALC) < 1,000 lymphocytes per microliter as determined by the complete blood count (CBC) differential analysis.

No current therapy exists for the regeneration and proliferation of the most important immune cells in the blood compartment responsible for cytotoxicity of tumor cells, the lymphocytes. Expanded access of NAI for the treatment of lymphopenia addresses an unmet medical need, since no therapy is currently approved to reverse a low lymphocyte count and maintain lymphocytes within the normal range. By offering patients the ability to treat lymphopenia, the potential exists of increasing overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Adult patients with solid tumors who progressed on standard-of-care treatment chemotherapy and/or immunotherapy and/or radiation therapy requiring second line or greater standard-of-care treatment with:

   * Chemotherapy and/or
   * Radiation therapy and/or
   * Immune checkpoint inhibitor therapy and/or any therapy investigator deems appropriate at that institution
3. Lymphocyte status meeting ONE of these conditions:

   * Baseline absolute lymphocyte count (ALC) <1,500 cells/μL (mild lymphopenia) prior to treatment initiation in first line therapy or ALC <1000 cells/μL (severe lymphopenia) during and or following progression after first line therapy
   * Anticipated treatment-induced lymphopenia (ALC reduction ≥20% from baseline based on reduction during first line therapy)
   * Persistent lymphopenia (ALC <1000 cells/μL for >2 months during first line therapy treatment)

Exclusion Criteria:

1. Active uncontrolled autoimmune disease requiring immunosuppression
2. Participants with liquid tumors
3. Concurrent solid organ transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon - Shiong Institute for Medicine, El Segundo, California, United States